CLINICAL TRIAL: NCT06779864
Title: Molecular Characteristics of Hepatitis B Virus Integration, Mutation, and Drug Resistance
Acronym: HBV IMDR
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Chief Physician, Beijing Friendship Hospital
Other Study IDs: 2023YFC2306903
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Hepatitis B
Keywords: HBV; HBV Mutation; HBV Integration; HBV Resistance
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum; Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antiviral treatment chronic hepatitis B cohort
- Hepatitis B patients in cross-sectional epidemiological survey cohort

SUMMARY:
Patients with a confirmed diagnosis of chronic hepatitis B (CHB) who have complete clinical data and retained blood or liver tissue samples will be enrolled. All patients will be grouped based on cohort sources: the Antiviral Treatment Cohort and the Cross-Sectional Epidemiological Survey Cohort.

Patients in the Antiviral Treatment Cohort have received antiviral treatment and are followed every six months. During follow-up, HBV-related endpoint events, including cirrhosis decompensations (such as ascites, esophageal variceal bleeding, and hepatic encephalopathy), hepatocellular carcinoma (HCC), liver transplantation, and liver-related death, will be collected.

In the Cross-Sectional Epidemiological Survey Cohort, clinical data will be collected at a single time point, with some patients not receiving antiviral treatment.

In both cohorts, retained blood and liver tissue samples will be used to further analyze HBV genotypes, viral integration, drug resistance, and the molecular characteristics of mutations.

Finally, a detailed description will be provided regarding the correlation between these HBV genetic molecular features and demographic distribution, clinical phases, and various clinical outcome events.

DETAILED DESCRIPTION:
To identify HBV genotypes, viral integration, drug resistance, and molecular characteristics of mutations associated with clinical immune phases and different clinical outcome events based on a representative hepatitis B clinical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatitis B surface antigen positive.
* Patients who have complete demographic information, clinical data and retained blood samples or liver tissue samples

Exclusion Criteria:

* Subject who without blood samples or liver tissue samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis B surface antigen positive, who have complete clinical data and retained blood samples or liver tissue samples.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in hepatitis B virus integration sites and count under antiviral treatment | Testing of previously collected samples within the time frame of 2015 to 2023

SECONDARY OUTCOMES:
Hepatitis B virus variants related to drug resistance under antiviral treatment | Testing of previously collected samples within the time frame of 2015 to 2023
Genetic mutations in Hepatitis B virus across different regions and populations. | Testing of previously collected samples within the time frame of 2014 to 2023
Genetic mutations in Hepatitis B virus related to different stages of disease progression | Testing of previously collected samples within the time frame of 2015 to 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No